CLINICAL TRIAL: NCT00929123
Title: Mechanisms of Neural Mobilization in the Treatment of Chronic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT002796 (NIH); R21AT002796 (NIH); R21AT002796-01A1 (NIH)
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: manual therapy; carpal tunnel syndrome; central sensitization
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- neural mobilization (Experimental): manual therapy technique known to directly stress the median nerve
  Interventions: Procedure: neural mobilization
- sham neural mobilization (Placebo Comparator): manual therapy technique known to directly stress the median nerve without any stimulation.
  Interventions: Procedure: sham neural mobilization
- Healthy Controls (Active Comparator): People without carpal tunnel syndrome for comparison
  Interventions: Other: healthy controls

INTERVENTIONS:
Procedure: neural mobilization — manual therapy technique known to directly stress the median nerve
  Other Names: upper limb tension test with median nerve bias
  Arms: neural mobilization
Procedure: sham neural mobilization — sham technique mimicking the neural mobilization which is not specific to the median nerve
  Arms: sham neural mobilization
Other: healthy controls — People without carpal tunnel syndrome for comparison
  Arms: Healthy Controls

SUMMARY:
The purpose of this study was to determine the effect of a manual therapy technique (neural mobilization) on measures of clinical pain and function, experimental pain sensitivity, and on the function of the median nerve in individuals with carpal tunnel syndrome. The investigators hypothesized that individuals receiving a neural mobilization technique known to directly stress the median nerve would demonstrate greater improvements in clinical pain and function, experimental pain sensitivity, and median nerve function than those receiving a sham technique.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* signs and symptoms of carpal tunnel syndrome for greater than 12 weeks

Exclusion Criteria:

* non english speaking
* prior surgery for carpal tunnel syndrome
* systemic condition known to affect sensation
* chronic pain condition other than carpal tunnel syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
thermal and pressure pain sensitivity | immediate effect

SECONDARY OUTCOMES:
grip strength | 3 weeks
wrist range of motion | 3 weeks
clinical pain | 3 weeks
self report of disability | 3 weeks
median nerve function | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z George, PhD, Principal Investigator — University of Florida Department of Physical Therapy
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Bialosky JE, Bishop MD, Price DD, Robinson ME, Vincent KR, George SZ. A randomized sham-controlled trial of a neurodynamic technique in the treatment of carpal tunnel syndrome. J Orthop Sports Phys Ther. 2009 Oct;39(10):709-23. doi: 10.2519/jospt.2009.3117. PMID 19801812
- [Result] Bialosky JE, Bishop MD, Robinson ME, Price DD, George SZ. Heightened pain sensitivity in individuals with signs and symptoms of carpal tunnel syndrome and the relationship to clinical outcomes following a manual therapy intervention. Man Ther. 2011 Dec;16(6):602-8. doi: 10.1016/j.math.2011.06.003. Epub 2011 Jul 20. PMID 21764354
- [Result] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342